CLINICAL TRIAL: NCT02490904
Title: Double-blind Placebo-Controlled Randomized Clinical Trial of Mineralocorticoid Receptor Blockade With Eplerenone After Renal Transplantation : Effect on Graft Function at 3 Months.
Brief Title: Eplerenone in Patients Undergoing REnal Transplant (EPURE TRANSPLANT)
Acronym: EPURE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Study chair, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-000956-29
Record Dates: First submitted 2015-07-01; First posted 2015-07-07 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: End-stage Renal Disease
Keywords: Kidney transplantation; Eplerenone
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone group (Experimental): Eplerenone administration within 2 hours prior to patient departure to the operating room and for 4 days after kidney transplantation.
  Interventions: Drug: Eplerenone
- Placebo group (Placebo Comparator): Placebo administration within 2 hours prior to patient departure to the operatingroom and for 4 days after kidney transplantation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — Double-blinded Eplerenone administered for 4 days at 25mg every 12 hours
  Arms: Eplerenone group
Drug: Placebo — Double-blinded Placebo administered for 4 days at 25mg every 12 hours
  Arms: Placebo group

SUMMARY:
Assess the impact of eplerenone (initiated within 2 hours prior to patient departure to the operating room and administered for 4 days during the post-operative period) on graft function evaluated by the measurement of glomerular filtration rate at 3 months - variable strongly associated with long-term graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Informed consent
* Candidate for a single or a dual kidney transplantation from an expanded criteria deceased donor ( 60 years or older or age between 50 and 59 with 2 of the 3 following criteria: cardiovascular death, history of hypertension, serum creatinine above 130µmol/L), regardless of machine perfusion and graft rank
* Chronic hemodialysis
* Affiliated to a social security system

Exclusion Criteria:

* Multiple organ transplantation (kidney and liver, kidney and heart, kidney and pancreas, kidney and lung, kidney and intestine)
* Patient receiving a graft from a donor under mineralocorticoid receptor antagonist treatment (spironolactone or eplerenone)
* Peritoneal dialysis
* Preemptive transplantation
* Hypersensitivity or known allergy to Eplerenone or one of its excipients
* Patients with severe hepatic insufficiency (class Child-Pugh C)
* Patient receiving powerful CYP3A4 inhibitors (for example itraconazole, ketoconazole, ritonavir, nelfinavir, clarithromycin, telithromycyn and nefazodone)
* Hypersensitivity or known allergy to iodinated contrast agents (iohexol)
* Demonstrated thyrotoxicosis
* Hypersensitivity to lactose
* HLA desensitization prior to renal transplantation
* Pregnant woman or woman without effective contraception
* Patient under judicial protection
* Patient under legal guardianship
* Participation in another biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2016-10-19 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Iohexol clearance | 3 months
  Graft function at 3 months evaluated by GFR using iohexol clearance

SECONDARY OUTCOMES:
Proportion of dialysis dependency | 3 months
Proportion of patients presenting a delayed graft function | 7 days post transplantation
  The proportion of patients with a delayed graft function defined by the need for one or more dialysis sessions during the 7 days following transplantation
24-hour proteinuria | 3 months
Occurrence of hyperkalemia > 6 mmol/l | 7 days post transplant
Length of initial hospital stay | 1 month
  between transplantation and discharge
Proportion of patients alive | 3 months 1 year, 3 years, 10 years
  vital status collected through the national database of organ recipients
serum creatinine | 3 months 1 year, 3 years, 10 years
  using the enzymatic method
glomerular filtration rate | 3 months 1 year, 3 years, 10 years
  estimation using the CKD-EPI formula (in mL/min/1.73m2)
Proportion of patients with immediate renal recovery, | 7 days post transplant
  The proportion of patients with an immediate renal recovery is defined by a serum creatinine lower than 30 mg/L at 7 days post-transplant
Iohexol clearance < 30 mL/min/1,73m² | 3 months
24-hour microalbuminuria | 3 months
Proportion of patients with a slow renal recovery | 7 days post transplant
  The proportion of patients with slow renal recovery is defined by serum creatinine above 30 mg/L at 7 days post-transplant without the need for dialysis
Proportion of patients with biopsy-proven acute rejection | 3 months post transplant
  Proportion of patients with biopsy-proven acute rejection in the first three month after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric JAISSER, MD, Principal Investigator — CHRU de Nancy; Sophie GIRERD, MD, Study Chair — CHRU de NANCY; Nicolas GIRERD, MD, PhD, Study Chair — CHRU de Nancy; Luc FRIMAT, MD, PhD, Study Chair — CHRU de Nancy; Patrick ROSSIGNOL, MD, PhD, Study Chair — CHRU de Nancy
Locations (7):
- France (7):
  - CHRU Besançon, Besançon
  - CHU Brest, Brest
  - CHU Dijon- Hôpital Bocage Central, Dijon
  - CHRU de Nancy, Nancy
  - CHU Reims-Hôpital Maison Blanche, Reims
  - CHU Saint Etienne, Saint-Etienne
  - NHC -CHRU Strasbourg, Strasbourg

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138
- [Derived] Girerd S, Frimat L, Ducloux D, Le Meur Y, Mariat C, Moulin B, Mousson C, Rieu P, Dali-Youcef N, Merckle L, Lepage X, Rossignol P, Girerd N, Jaisser F. EPURE Transplant (Eplerenone in Patients Undergoing Renal Transplant) study: study protocol for a randomized controlled trial. Trials. 2018 Oct 30;19(1):595. doi: 10.1186/s13063-018-2956-1. PMID 30376884

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT02490904/SAP_000.pdf